CLINICAL TRIAL: NCT06360978
Title: Efficacy and Toxicity of Docetaxel as a Radiosenstizer in Head and Neck Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Rehab Osama Abdelmaboud, assistant lecturer, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: docetaxel as a radiosenstizer
Record Dates: First submitted 2024-03-29; First posted 2024-04-11 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Docetaxel — Our patients will receive docetaxel (15 mg per meter squared) once weekly concurrently with radiotherapy.

SUMMARY:
Head and neck cancer (HNC) is the seventh most common cancer globally, accounting for more than 660,000 new cases and 325,000 deaths annually. The overall incidence of HNC continues to rise, with a predicted 30% increase annually by 2030., this increase has been recorded across both developed and developing countries.

Approximately 90% of HNCs are squamous cell carcinoma . The major risk factors of head and neck squamous cell carcinoma (HNSCC) are tobacco and heavy alcohol use and human papillomavirus infection . There has been a significant decline in smoking in high-income countries during the last few decades, which has led to a sharp decline in smoking related HNSCC . While increase in global incidence of human papillomavirus (HPV)-associated or positive (+) HNSCC Head and neck squamous cell carcinoma (HNSCC) is a highly challenging cancer, despite the advancements in treatment, the overall prognosis for HNSCC remains poor, with a five-year survival rate of around 50%.

Chemoradiation is one of the treatment options for locally advanced head and neck cancers, the drug of choice for radiosensitization is cisplatin Although cisplatin-based chemoradiotherapy (CRT) is the standard of care for locally advanced head and neck squamous cell carcinoma (LAHNSCC), cisplatin is contraindicated in many patients because of age, diminished renal functions and hearing loss so docetaxel studied as an alternative radiosensitizer in this group.

The addition of docetaxel to radiation improved DFS and OS in cisplatin-ineligible patients with LAHNSCC.

DETAILED DESCRIPTION:
History: age, gender, comorbidities and risk factors.

Baseline evaluation of the patients:

CT or MRI head and neck Endoscopy and biopsy will be taken. Laboratory: CBC, renal functions and liver functions Nutritional assessment Audiogram as baseline assessment Dental assessment

Our patients will receive docetaxel (15 mg per meter squared) once weekly concurrently with radiotherapy.

Follow up of the patient during the course of treatment including evaluation of the patients weekly to assess the adverse events in the form of skin toxicity, mucositis, neutropenia and renal function affection.

Follow up after finishing the course of treatment. After 6 to 8 weeks the patient will be evaluated with CT or MRI head and neck and endoscopy Then every three month we will evaluate the patient as regarding the quality of life and late toxicity up to 2 years

ELIGIBILITY:
Inclusion Criteria:

* Patients above 18 years
* Pathologically proven of squamous cell carcinoma
* Patients with locally advanced disease (T3, T4)(N positive)
* Patients eligible for radiotherapy

Exclusion Criteria:

* Patients with metastatic disease
* Patients with second primary cancer
* Patients ineligible for radiotherapy

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
progression free survival | 2 years
  Progression free survival defined as the average length of time after the start of treatment in which a person is alive and their cancer does not grow or spread

SECONDARY OUTCOMES:
incidence of treatment adverse events | 2 years
  evaluation of any adverse events will be occurred during treatment and 2 years after
Overall survival (OS) | 2 years
  Overall survival defined as the average length of time patients are alive after diagnosis or the start of treatment.

IPD SHARING:
Plan to Share IPD: No